CLINICAL TRIAL: NCT05872776
Title: A Multi Center Randomized, Double Blinded, Sham Controlled, Clinical Study Aimed to Determine the Efficacy of CardiaCare™ RR2 Home-care Neuromodulation System in Reducing Atrial Fibrillation Burden and Symptoms in Paroxysmal AF Patients
Brief Title: BEAT AF - Braking Ectopic Atrial Trends In Atrial Fibrillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziv HealthCare Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAR-POC-02
Record Dates: First submitted 2023-04-30; First posted 2023-05-24 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RR2 wearable home-care: active device (Active Comparator): Real stimulation with RR2 neuromodulation device
  Interventions: Device: Neuromodulation with RR2 device
- RR2 wearable home-care: sham control device (Sham Comparator): Mock sham stimulation with RR2 neuromodulation device
  Interventions: Device: Mock sham neuromodulation with sham RR2 device

INTERVENTIONS:
Device: Neuromodulation with RR2 device — non-invasive neuromodulation with RR2 device
  Arms: RR2 wearable home-care: active device
Device: Mock sham neuromodulation with sham RR2 device — Mock sham stimulation with RR2 device
  Arms: RR2 wearable home-care: sham control device

SUMMARY:
Paroxysmal AF subjects with a documented ECG event of AF will be recruited to the study To assess the efficacy of CardiaCare™ RR2 wearable home-care neuromodulation system in reducing AF burden and symptoms in Paroxysmal AF patients

DETAILED DESCRIPTION:
After screening for 14 days with a continuous ECG monitoring device, eligible patients will be randomized to either active treatment or a sham treatment groups. For a treatment period of 12 weeks, patients will be prompted to self-conduct neuromodulation sessions based on: a. predetermined treatment regimen plus b. a detection algorithm. In addition, participants will measure at home, daily 2 min ECG's with the RR2 system two times a day and when feeling symptoms suspected as AF/AT/SVT or PAC's.

After 10 weeks of treatment patients will be requested to wear an ECG patch continuously for an additional period of 14 days.

Overall patients will participate in the study for 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-85 years with history of documented paroxysmal (<7 days) atrial fibrillation
* AF Burden (% time in AF) of more than 0.5% and less than 25% as evident by a continuous 14 days ECG recording at baseline (at minimum 168 hours)
* Ability and willingness to sign an informed consent form
* Ability and willingness to use CardiaCare home care device and ECG chest patch and has an available smart phone
* Known symptomatic AF event over the recent 3 months
* Willing not to change the antiarrhythmic treatment

Exclusion Criteria:

* Hemodynamic instability (systolic blood pressure <100mmHg or heart rate>170 bpm at Baseline) during recruitment visit
* Known history or current diagnosis of atrial flutter
* An active myocardial infarction evident from ECG
* Recent stroke or myocardial infarction (<6 months)
* History of sick sinus syndrome 2nd or 3rd degree AV block, bifascicular block or prolonged (PR>300ms) 1st degree AV block
* Unilateral or bilateral vagotomy
* History of persistent AF with documented AF episodes of >7 days
* Significant valvular disorder (i.e., prosthetic valve or hemodynamically relevant valvular diseases or valvular AF)
* History of Impaired systolic function with EF<40 % or NY Class III or IV heart failure classification
* Dilatated left atria with a diameter > 50mm as evident by an echocardiogram
* Currently enrolled in another study
* Recurrent vaso-vagal syncopal episodes
* Pregnancy or breast feeding
* Pacemaker or CRTD or any implanted electrical stimulating device
* History of epilepsy or seizures
* Peripheral neuropathy or dermatological condition affecting the tested upper extremity area
* Unsuitable for participating in the study according to attending physician

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change in AF burden | 14 weeks
  Defined as % of time in AF, during screening period compared to end of treatment period.

SECONDARY OUTCOMES:
AF burden defined as the total number of AF events during screening period compared to end of treatment period. | 14 weeks
AF burden defined as the total number of symptomatic AF events during screening period compared to end of treatment period | 14 weeks
Change from baseline compared to end of treatment period in Life quality & symptoms as assessed by AF AFEQT(from 0-poor to 100-great), EHRA Score (from I-no symptoms to IV-disabling symptoms) and SF36 questionnaires (form 0-worst to 100-best) | 14 weeks
Number of AF episodes lasting 6 hours or longer in the treatment arm compared to the sham control | 14 weeks
Group change in acute reduction of PAC (number of PACs in 2 minute ECG) compared before and immediately after neuromodulation sessions | 14 weeks
Mean group change in ATA (Atrial Tachyarrhythmias, score form 0 to 6)/ PAC ( Premature Atrial Contractions, number of PACs in 2 minute ECG ) burden from Screening period to End of treatment period | 14 weeks
Proportion of patients with 20% change in ATA /PAC (Premature Atrial Contractions, measured 14 days continuance ECG) burden | 14 weeks
Mean group change in acute reduction of PAC (number of PACs in 2 minute ECG) compared before to up to 1 hour after each neuromodulation session | 14 weeks
Adherence: proportion of executed Vs. planned self-treatments delivered by each patient throughout the treatment period | 14 weeks
Safety- number of AE | 14 weeks
  number and severity of adverse event
Patient satisfaction and preferences as assessed by patient centric (0-none to 10-worst) & usability questionnaires (1-strongly disagree to 5-strongly agree) | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Chorin, MD, Principal Investigator — Tel Aviv Souraski Medical Center, Department of Cardiology
Locations (2):
- Israel (2):
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Clalit Health Services (HMO), Tel Aviv

IPD SHARING:
Plan to Share IPD: No